CLINICAL TRIAL: NCT03806608
Title: Clinical and Radiographic Evaluation of Marginal Bone Changes Around Platform-switching Implants Placed in Crestal or Subcrestal Positions: a Randomized Controlled Clinical Trial
Brief Title: Evaluation of MBL Around Implants Placed in Crestal or Subcrestal Positions: a RCT
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Sun Yat-sen University (Other)
Responsible Party: Principal Investigator, Baoxin Huang, Principle Investigator, Sun Yat-sen University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: Baoxin Huang Depth
Record Dates: First submitted 2019-01-14; First posted 2019-01-16 (Actual); Last update posted 2022-04-20 (Actual); Status verified 2022-04

CONDITIONS: Jaw, Edentulous; Partial Edentulism
Keywords: Marginal Bone Loss; Implant depth; Crestal or Subcrestal
MeSH Terms: conditions — Jaw, Edentulous

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Crestal (Experimental): Implants were placed with the implant-abutment interface(IAI) at the level of the the alveolar ridge
  Interventions: Procedure: Crestal
- Subcrestal (Experimental): Implants were placed with the implant-abutment interface(IAI) 1 mm below the level of the alveolar ridge
  Interventions: Procedure: Subcrestal

INTERVENTIONS:
Procedure: Crestal — Subjects will be included with the absence of 2-4 teeth in the posterior region of the maxilla or mandibular. Twenty patients will be recruited. Two implant placement depths, equicrestal and subcrestal, were randomly assigned to two sites of each patient with a predefined randomization tables (one crestal implant and one subcrestal implant).
  Arms: Crestal
Procedure: Subcrestal — Subjects will be included with the absence of 2-4 teeth in the posterior region of the maxilla or mandibular. Twenty patients will be recruited. Two implant placement depths, equicrestal and subcrestal, were randomly assigned to two sites of each patient with a predefined randomization tables (one crestal implant and one subcrestal implant).
  Arms: Subcrestal

SUMMARY:
The objective of this randomized controlled trial is to evaluate changes in marginal bone levels and soft tissue dimensions around implants placed with the IAI at different positions in relation to the alveolar crest

DETAILED DESCRIPTION:
The objective of this randomized controlled trial is to evaluate changes in marginal bone levels and soft tissue dimensions around implants placed with the IAI at different positions in relation to the alveolar crest. Subjects will be included with the absence of 2-4 teeth in the posterior region of the maxilla or mandibular. Twenty patients will be recruited. Two implant placement depths, equicrestal and subcrestal, were randomly assigned to two sites of each patient with a predefined randomization tables (one crestal implant and one subcrestal implant). Patients will be recalled for oral hygiene maintenance and prosthetic controls at 1year, 3 years, 5 years after final restoration.

ELIGIBILITY:
Inclusion Criteria:

1. Absence of 2-4 teeth in the posterior region of the maxilla or mandibular;
2. Bone volume sufficient for implants with 4.1-mm size and 8- to 12-mm height and with no need for hard or soft tissue augmentation for implant treatment;
3. Periodontally healthy.

Exclusion Criteria:

1. Systemic diseases that may affect bone and soft tissue healing, such as diabetes, osteoporosis, Paget's disease, and patients with cancer;
2. Uncontrolled periodontal disease or poor oral health with neither good nor adequate plaque control;
3. Parafunctional habits, such as the grinding or clenching of teeth;
4. Smoking habit (more than 10 cigarettes per day);
5. Pregnancy and breastfeeding.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2019-04-17 (Actual); Primary Completion 2026-05 (Estimated); Study Completion 2026-05 (Estimated)

PRIMARY OUTCOMES:
Marginal bone loss(MBL) | Change from baseline up to 5 years after implantation
  Baseline will be recorded at the time of implantation. Margin bone loss(MBL) will be recorded at 0 day, 4 months, 1 year and 3 years after implant placement.

SECONDARY OUTCOMES:
Cumulative survival rate (CSR) | Up to 5 years after final restoration
  Cumulative survival rate will be assessed at final restoration, 1 year, 3 years, 5 years after final restoration
Pocket probing depth (PPD) | Up to 5 years after final restoration
  Pocket probing depth will be assessed at 1 year, 3 years, 5 years after final restoration
Plaque index (PI) | Up to 5 years after final restoration
  Plaque index will be assessed at 1 year, 3 years, 5 years after final restoration
Bleeding on probing (BOP) | Up to 5 years after final restoration
  Bleeding on probing will be assessed at 1 year, 3 years, 5 years after final restoration

CONTACTS AND LOCATIONS:
Overall Officials: Baoxin Huang, PhD, Principal Investigator — Sun Yat-sen Unniversity
Locations (1):
- Guanghua School of Stomatology,Hospital of Stomatology,Sun Yat-Sen University, Guangzhou, Guangdong, China

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Huang B, Meng H, Zhu W, Witek L, Tovar N, Coelho PG. Influence of placement depth on bone remodeling around tapered internal connection implants: a histologic study in dogs. Clin Oral Implants Res. 2015 Aug;26(8):942-949. doi: 10.1111/clr.12384. Epub 2014 Apr 10. PMID 24720447
- [Background] Huang B, Meng H, Piao M, Xu L, Zhang L, Zhu W. Influence of placement depth on bone remodeling around tapered internal connection implant: a clinical and radiographic study in dogs. J Periodontol. 2012 Sep;83(9):1164-71. doi: 10.1902/jop.2012.110617. Epub 2012 Jan 5. PMID 22220773
- [Background] Koutouzis T, Neiva R, Nonhoff J, Lundgren T. Placement of implants with platform-switched Morse taper connections with the implant-abutment interface at different levels in relation to the alveolar crest: a short-term (1-year) randomized prospective controlled clinical trial. Int J Oral Maxillofac Implants. 2013 Nov-Dec;28(6):1553-63. doi: 10.11607/jomi.3184. PMID 24278924
- [Background] Valles C, Rodriguez-Ciurana X, Clementini M, Baglivo M, Paniagua B, Nart J. Influence of subcrestal implant placement compared with equicrestal position on the peri-implant hard and soft tissues around platform-switched implants: a systematic review and meta-analysis. Clin Oral Investig. 2018 Mar;22(2):555-570. doi: 10.1007/s00784-017-2301-1. Epub 2018 Jan 8. PMID 29313133